CLINICAL TRIAL: NCT02321540
Title: A Phase I/II Study of Ibrutinib in Previously Treated Epidermal Growth Factor Receptor (EGFR) Mutant Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0602; NCI-2015-00124 (Registry Identifier: NCI CTRP); 1R01CA190628 (NIH)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; NSCLC; Epidermal growth factor receptor mutations; EGFR; Recurrent non-small cell lung cancer; Ibrutinib; PCI-32765; Imbruvica
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Participants in Part 1 receive dose level of Ibrutinib depending on study joined. First group of participants receive lowest dose level of Ibrutinib. Each new group receives a higher dose of Ibrutinib than the group before it, if no intolerable side effects were seen. This continues until highest tolerable dose of Ibrutinib is found.
  Participants in Part 2 receive Ibrutinib at highest dose that was tolerated in Part 1 or 840 mg daily.
  Starting level of Ibrutinib: 560 mg by mouth daily in a 28 day cycle.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Part 1 Starting level of Ibrutinib: 560 mg by mouth daily in a 28 day cycle.
  Part 2 Starting level of Ibrutinib: Maximum tolerated dose from Part 1 or 840 mg daily.
  Other Names: PCI-32765; Imbruvica

SUMMARY:
The goal of Part 1 of this clinical research study is to find the highest dose of (Imbruvica) ibrutinib that can be given to patients with non-small cell lung cancer (NSCLC). The goal of Part 2 of this clinical research study is to learn if the dose of ibrutinib found in Part 1 can help to control the disease.

The safety of this drug will also be studied in both parts of the study.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of up to 6 participants will be enrolled in Part 1 of the study, and up to19 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of ibrutinib you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of ibrutinib. Each new group will receive a higher dose of ibrutinib than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ibrutinib is found.

If you are enrolled in Part 2, you will receive ibrutinib at the highest dose that was tolerated in Part 1.

Study Drug Administration:

You will take ibrutinib pills 1 time each day, at about the same time every day. You may take your dose of ibrutinib with or without food.

Study Visits:

Each cycle is 4 weeks.

On Day 1 of all cycles:

* You will have a physical exam
* Blood (about 3 teaspoons) will be drawn for routine tests.
* On Cycle 2 only, blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing before your dose and then 4 more times over the next 6 hours after your dose. PK testing measure the amount of study drug in the body at different timepoints.
* If you the doctor thinks it is needed, blood (about ½ teaspoon) or urine will be collected for pregnancy testing.

Every 8 weeks, you will have a CT, MRI, or x-ray to check the status of the disease. You will have the same type of scan performed as you did at screening.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Dosing Visit:

About 30 days after your last dose of study drug:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* If you the doctor thinks it is needed, blood (about ½ teaspoon) or urine will be collected for pregnancy testing.

Follow Up Visits:

Every 6 months you will be asked to come into the clinic or you will be called by a member of the study staff to ask how you are doing and if you have started any new anti-cancer treatments. If you are called, it should take about 10 minutes.

This is an investigational study. Ibrutinib is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia (CLL) and mantle cell lymphoma (MCL). It is considered investigational to use this drug to treat NSCLC. The study doctor can explain how the study drug is designed to work.

Up to 43 participants will be enrolled on this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed stage IV non-small cell lung cancer, or recurrent non-small cell lung cancer which is not amenable to curative intent therapy.
2. Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 criteria
3. For EGFR mutant cohort, patients must have: a) Documented EGFR mutation by Clinical Laboratory Improvement Amendments (CLIA)-certified test b) Documented disease progression on treatment with erlotinib, gefitinib, afatinib, or other EGFR-targeted tyrosine kinase inhibitor c) Tissue available from a biopsy or surgical procedure performed after progression on an EGFR targeted tyrosine kinase inhibitor. If tissue is not available, the patient must have biopsy accessible disease and must be willing to undergo a biopsy.
4. For HER2 mutant cohort, patients must have: a) Documented EGFR mutation by CLIA-certified test b)Documented disease progression on treatment with erlotinib, gefitinib, afatinib, or other EGFR-targeted tyrosine kinase inhibitor c)Tissue available following progression on most recent systemic therapy. If tissue is not available, the patient must have biopsy accessible disease and must be willing to undergo a biopsy.
5. Age >/=18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status </=2
7. Ability to take pills by mouth
8. Patients must have normal organ and marrow function as defined: leukocytes >/= 3,000/mcL; absolute neutrophil count >/= 1,500/mcL; hemoglobin >/= 9 g/dL; total bilirubin </= 1.5 x institutional upper limit of normal (ULN); AST(SGOT)/ALT(SGPT) </= 2.5 × ULN or </= 5 x ULN if metastases to the liver; creatinine clearance >/= 45 mL/min
9. Patients with asymptomatic brain metastases are allowed, as long as they are stable and do not require treatment with anticonvulsants or escalating doses of steroids. Maximum daily dose of steroids should be prednisone 20 mg or equivalent. Radiation therapy for brain metastases must be completed at least 14 days prior to treatment on protocol
10. The effects of ibrutinib on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use highly effective contraception (if using hormonal birth control must add a second barrier method; abstinence) prior to study entry, for the duration of study participation as well as for at least 1 month after the last dose of ibrutinib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use highly effective contraception prior to the study, for the duration of study participation and 3 months after completion of ibrutinib administration.
11. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients who have received EGFR tyrosine kinase inhibitors within 72 hours of initiation of study treatment, or treatment with other anti-cancer agents within 21 days of study treatment
2. Prior treatment with ibrutinib
3. Known hypersensitivity to ibrutinib
4. Concurrent use of agents that strongly inhibit or induce CYP3A unless use is approved by the medical monitor
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Pregnant and nursing women
7. Patients with a history of another active malignancy within the past two years, with the exception of non-melanoma cutaneous malignancy, cervical carcinoma in situ, or ductal carcinoma in situ which has been successfully treated with curative intent therapy
8. Any gastrointestinal disorder expected to limit absorption of ibrutinib
9. Treatment with warfarin or other vitamin K antagonist. Patients with using warfarin who switch to another form of anticoagulation will be eligible
10. Patients with persistent and uncontrolled atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Heymach, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib Dose Level 0: Participants received Ibrutinib at dose level 0 (560 mg PO daily) on a continuous basis on 28 day cycles.
- Ibrutinib Dose Level 1: Participants received dose level 1 (840 mg PO daily) on a continuous basis on 28 day cycles.
Period: Overall Study
Arm/Group | Ibrutinib Dose Level 0 | Ibrutinib Dose Level 1
Started | 3 | 10
Completed | 0 | 0
Not Completed | 3 | 10
Not completed — Death | 0 | 1
Not completed — Progression | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Ibrutinib Dose Level 0: Participants received Ibrutinib at dose level 0 (560 mg PO daily on a continuous basis on 28 day cycles.
- Ibrutinib Dose Level 1: Participants received Ibrutinib dose level 1 (840 mg PO daily) on a continuous basis on 28 day cycles.
- Total: Total of all reporting groups
Arm/Group | Ibrutinib Dose Level 0 | Ibrutinib Dose Level 1 | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 6 | 6
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 12
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity (DLT) Observed During the Dose Escalation to Determine the Maximum Tolerated Dose (MTD)
Description: Number of DLT observed at dose levels 560 (starting dose) and 840 mg PO daily to determine the MTD using the 3+3 design.
Time Frame: First cycle of 28 days
Population: 12 patients were evaluable for overall response rate; 1 patient who received 840 mg PO daily was inevaluable due to death prior to first response assessment after start of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Ibrutinib Dose Level 0 (560mg): Participants received Ibrutinib at dose level 0 (560 mg PO daily) on a continuous basis on 28 day cycles.
- Ibrutinib Dose Level 1 (840mg): Participants received Ibrutinib at dose level 1 (840 mg PO daily) on a continuous basis on 28 day cycles.
Arm/Group | Ibrutinib Dose Level 0 (560mg) | Ibrutinib Dose Level 1 (840mg)
Number analyzed (Participants) | 3 | 10
Participants | 0 | 0

2. Primary Outcome: Overall Response Rate in Patients With EGFR Mutations Using RECIST
Description: Complete response and partial resopnse rate RECIST 1.1 criteria The response was evaluated after two cycles of therapy and every 8 weeks until the first date that recurrent or progressive disease is objectively documented, up to 2 years.
Time Frame: after two cycles of therapy and every 8 weeks, up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Ibrutinib Dose Level 0 (560mg): Participants received ibrutinib at dose level 0 (560 mg daily).
- Ibrutinib Dose Level 1 (840mg): Participants received Ibrutinib at dose level 1 ( 840 mg PO daily).
Arm/Group | Ibrutinib Dose Level 0 (560mg) | Ibrutinib Dose Level 1 (840mg)
Number analyzed (Participants) | 3 | 9
Participants | 3 | 9

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the duration of time from start of treatment to time of progression or death.
Time Frame: from start of treatment to time of progression or death, up to 2 years
Population: 13 patients were followed up 12 patients were evaluable for disease control rate, duration of response and Response rate in patients with HER2 mutant non-small cell lung cancer; 1 patient who received 840 mg PO daily was inevaluable due to death prior to first response assessment after start of treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ibrutinib Dose Level 0 (560mg): Participants received Ibrutinib at dose level 0 (560 mg PO daily, starting dose) and dose level 1 (840 mg PO daily).
- Ibrutinib Dose Level 1 (840mg): Participants received Ibrutinib at dose level 1 (840 mg PO daily).
Arm/Group | Ibrutinib Dose Level 0 (560mg) | Ibrutinib Dose Level 1 (840mg)
Number analyzed (Participants) | 3 | 10
months | 13.6 [6.4 to 14.4] | 10.3 [0.67 to 16.0]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: from start of treatment to time progression or death, whichever occurs first, up to 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ibrutinib Dose Level 0 (560mg): Participants received Ibrutinib at dose level 0 (560 mg PO daily, starting dose).
- Ibrutinib Dose Level 1 (840mg): Participants received Ibrutinib at dose level 1 (840 mg PO daily, starting dose).
Arm/Group | Ibrutinib Dose Level 0 (560mg) | Ibrutinib Dose Level 1 (840mg)
Number analyzed (Participants) | 3 | 10
months | 1.83 [1.70 to 1.87] | 1.75 [0.67 to 2.00]

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication, up to 2 years
Groups:
- Ibrutinib at Dose Level 0 (560 PO Daily).: Participants received Ibrutinib at dose level 0 (560 mg PO daily)
- Ibrutinib at Dose Level 1 (840 PO Daily).: Participants received Ibrutinib at dose level 1 (840 mg PO daily)
Arm/Group | Ibrutinib at Dose Level 0 (560 PO Daily). | Ibrutinib at Dose Level 1 (840 PO Daily).
All-Cause Mortality (participants affected / at risk) | 3/3 | 10/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/10
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib at Dose Level 0 (560 PO Daily). (N=3) | Ibrutinib at Dose Level 1 (840 PO Daily). (N=10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib at Dose Level 0 (560 PO Daily). (N=3) | Ibrutinib at Dose Level 1 (840 PO Daily). (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burning with urination (Infections and infestations) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Congestion of chest (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (7)
Decreased chloride (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (6)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (2)
Elevated UAWBC NCS (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Mild dry rash a little on chest and arms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash on legs and stomach (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) — Tenderness, right mid abdomen wall
Tightness of upper left lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine output decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (7)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02321540/Prot_SAP_000.pdf